CLINICAL TRIAL: NCT04621175
Title: Determining Optimal Energy Substrate to Enhance Postprandial Protein Kinetic Responses to Essential Amino Acid-enriched Whey During Energy Deficit
Brief Title: Effects of Essential Amino Acid-enriched Whey and Carbohydrate Co-ingestion on Protein Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: University of Arkansas (Other); Eastern Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20-14HC
Record Dates: First submitted 2020-08-24; First posted 2020-11-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-10

CONDITIONS: Energy Deficit
Keywords: whole-body protein turnover; muscle protein synthesis; protein kinetics
MeSH Terms: interventions — Carbohydrates; Excitatory Amino Acids

STUDY DESIGN:
Intervention Model Description: randomized, cross-sectional, longitudinal study
Who Masked: Participant, Investigator
Masking Description: double (participant and investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EAA+W & Carbohydrate: Balance (BAL) first, then Deficit (DEF) (Active Comparator): Participants will consume an essential amino acid plus whey (EAA+W) beverage with added Carbohydrate during energy balance (BAL) first, then again during energy deficit (DEF).
  Interventions: Dietary Supplement: EAA+W & Carbohydrate
- EAA+W & Carbohydrate: DEF first, then BAL (Active Comparator): Participants will consume an essential amino acid plus whey beverage with added Carbohydrate during energy deficit first, then again during energy balance.
  Interventions: Dietary Supplement: EAA+W & Carbohydrate
- EAA+W & EAA: BAL first, then DEF (Active Comparator): Participants will consume an essential amino acid (EAA) plus whey beverage with added EAA during energy balance first, then again during energy deficit.
  Interventions: Dietary Supplement: EAA+W & EAA
- EAA+W & EAA: DEF first, then BAL (Active Comparator): Participants will consume an essential amino acid (EAA) plus whey beverage with added EAA during energy deficit first, then again during energy balance.
  Interventions: Dietary Supplement: EAA+W & EAA

INTERVENTIONS:
Dietary Supplement: EAA+W & Carbohydrate — Essential amino acid plus whey beverage with added carbohydrate
  Arms: EAA+W & Carbohydrate: Balance (BAL) first, then Deficit (DEF); EAA+W & Carbohydrate: DEF first, then BAL
Dietary Supplement: EAA+W & EAA — Essential amino acid plus whey beverage with added essential amino acid
  Arms: EAA+W & EAA: BAL first, then DEF; EAA+W & EAA: DEF first, then BAL

SUMMARY:
Previous work conducted by the Investigators demonstrates that an essential amino acid(EAA)-enriched whey protein combination format is an efficient EAA/protein format to support enhanced whole-body protein balance and sustain muscle protein synthesis compared to isonitrogenous amounts of whey alone or a mixed-macronutrient meal. However, additional work is needed to optimize the formulation to ensure the best possible muscle and whole-body anabolic responses are achieved. This includes addressing the potential value of adding non-EAA/protein components to support energy demands. Providing additional non-protein energy to an EAA-enriched whey protein formulation may reduce the proportion of exogenous amino acids directed towards energy production thereby preserving its use for muscle protein synthesis. However, whether suppressing exogenous amino acid oxidation by providing additional carbohydrate allows for a greater muscle protein synthetic stimulus during moderate energy deficit (- 30% total energy requirements) is unknown. Therefore, this study will test the effects of EAA-enriched whey protein plus carbohydrate versus EAA-enriched whey plus additional EAA using a randomized, cross-sectional longitudinal study design.

DETAILED DESCRIPTION:
In this study the Investigators will test the effects of EAA-enriched whey protein plus carbohydrate versus EAA-enriched whey plus additional EAA using a randomized, cross-sectional longitudinal study design. Thirty healthy, functional and aerobic exercise trained adults will complete two, 5-d controlled feeding phases, one maintaining energy balance and one inducing energy deficit in random order and separated by at least a 7d washout period. The difference in post-exercise (whole-body exercise model) muscle protein synthesis and whole-body protein turnover between the study treatments will be determined the day after each 5-d controlled feeding phase. This design will test the following hypotheses: 1) The magnitude of post-exercise anabolic response to EAA-enriched whey protein plus carbohydrate are enhanced compared to EAA-enriched whey protein plus additional EAA during energy deficit; 2) Regardless of protein treatment, the magnitude of anabolic response will be reduced during energy deficit compared to energy balance.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30.0 kg/m2
* Weight stable in the past 2 months (± 2.27 kg)
* Healthy without evidence of chronic illness or musculoskeletal injury as determined by the USARIEM Office of Medical Support and Oversight (OMSO) or home duty station medical support
* Functional exercise (i.e., step ups, box jumps, body mass movements) and/or aerobic exercise trained defined by self-report as performing ≥ 2 sessions/wk for previous 6 months
* Willing to refrain from taking any nonsteroidal anti-inflammatory drugs (e.g., aspirin, Advil®, Aleve®, Naprosyn®), or any other aspirin-containing product for 10 days before the first ~8.5 hour laboratory day and at least 5 days after completing the last ~8.5 hour laboratory day
* Willing to refrain from alcohol, smoking any nicotine product (includes e-cigarettes), vaping, chewing tobacco, caffeine, and dietary supplements after the completing the baseline period until the end of the study
* Must obtain supervisor approval for federal civilian employees and non-HRV active duty military personnel working within the US Army Natick Soldier Systems Center
* Females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or able to provide documentation of oral/hormonal contraceptive use which contains low-dose estrogen/progesterone to maintain continuous levels throughout the 28-day cycle (i.e., no placebos)

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities, gastrointestinal disorders (e.g., kidney disease, diabetes, cardiovascular disease, etc.)
* Abnormal PT/PTT test or problems with blood clotting
* History of complications with lidocaine
* Present condition of alcoholism, anabolic steroids, or other substance abuse issues as assessed by OMSO
* Participation in blood donation within 8-wk of beginning the study
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test or self-report for breastfeeding will be obtained before body composition testing)
* Unwillingness or inability to consume study diets or foods provided due to personal preference, dietary restrictions, and/or food allergies
* Unwillingness to adhere to study physical restrictions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Whole-body Protein Balance | approximately 5.75 hours
  Whole-body net balance will be determined using stable-isotope methodologies
Whole-body Protein Synthesis | approximately 5.75 hours
  Whole-body protein synthesis will be determined using stable-isotope methodologies
Whole-body Protein Breakdown | approximately 5.75 hours
  Whole-body protein breakdown will be determined using stable-isotope methodologies
Muscle Protein Synthesis | approximately 5.75 hours
  Muscle protein synthesis will be determined using stable-isotope methodologies

CONTACTS AND LOCATIONS:
Overall Officials: Jess A Gwin, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwin JA, Robillard JT, Murphy NE, Carrigan CT, Wilson MA, Varanoske AN, Church DD, Ferrando AA, Pasiakos SM, Margolis LM. Elevated miR-194-5p Expression During Short-term Energy Deficit Attenuates Post-Exercise Muscle Protein Synthesis by Inhibiting Anabolic Signaling. J Nutr. 2026 Jan 27:101380. doi: 10.1016/j.tjnut.2026.101380. Online ahead of print. PMID 41611130
- [Derived] Gwin JA, Church DD, Allen JT, Wilson MA, Carrigan CT, Murphy NE, Varanoske AN, Margolis LM, Wolfe RR, Ferrando AA, Pasiakos SM. Consuming Whey Protein with Added Essential Amino Acids, Not Carbohydrate, Maintains Postexercise Anabolism While Underfed. Med Sci Sports Exerc. 2025 Jan 1;57(1):70-80. doi: 10.1249/MSS.0000000000003541. Epub 2024 Aug 23. PMID 39160756